CLINICAL TRIAL: NCT01026623
Title: Phase I/II Trial of Anti-IGF-IR Monoclonal Antibody IMC-A12 Plus mTOR Inhibitor Temsirolimus (CCI-779) in Metastatic Castration-Resistant Prostate Cancer (CRPC)
Brief Title: Cixutumumab and Temsirolimus in Treating Patients With Metastatic Prostate Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2011-01406; NCI-2011-01406 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000659064; 09-117; 09-117 (Other: Memorial Sloan-Kettering Cancer Center); 8147 (Other: CTEP); P30CA008748 (NIH); U01CA069856 (NIH)
Record Dates: First submitted 2009-12-03; First posted 2009-12-04 (Estimated); Results first posted 2019-06-17 (Actual); Last update posted 2019-06-17 (Actual); Status verified 2019-05

CONDITIONS: Hormone-Resistant Prostate Cancer; Prostate Adenocarcinoma; Recurrent Prostate Carcinoma; Stage IV Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — cixutumumab; temsirolimus; Sirolimus

ARMS (1):
- Treatment (cixutumumab, temsirolimus) (Experimental): Patients receive cixutumumab IV over 60-70 minutes and temsirolimus IV over 30 minutes on days 1, 8, 15, and 22. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: Cixutumumab; Other: Diagnostic Laboratory Biomarker Analysis; Drug: Temsirolimus

INTERVENTIONS:
Biological: Cixutumumab — Given IV
  Other Names: Anti-IGF-1R Recombinant Monoclonal Antibody IMC-A12; IMC-A12
Other: Diagnostic Laboratory Biomarker Analysis — Correlative studies
Drug: Temsirolimus — Given IV
  Other Names: CCI-779; CCI-779 Rapamycin Analog; Cell Cycle Inhibitor 779; Rapamycin Analog; Rapamycin Analog CCI-779; Torisel

SUMMARY:
This phase I/II trial is studying the side effects of giving cixutumumab together with temsirolimus and to see how well it works in treating patients with metastatic prostate cancer. Monoclonal antibodies, such as cixutumumab, can block tumor growth in different ways. Some block the ability of tumor cells to grow and spread. Others find tumor cells and help kill them or carry tumor-killing substances to them. Temsirolimus may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Giving cixutumumab together with temsirolimus may kill more tumor cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To confirm the safety and tolerability of IMC-A12 (cixutumumab) and temsirolimus using the recommended phase II dose level for advanced solid tumors in chemo-naive patients with metastatic castration-resistant prostate cancer and a rising prostate-specific antigen (PSA). (Phase I) II. To confirm the safety and tolerability of IMC-A12 and temsirolimus given on an every three weeks dosing schedule. (Phase I Extension) II. To determine the tumor response rate and/or composite time to progression (cTTP) for chemotherapy-naive patients with castration-resistant prostate cancer (CRPC) receiving the combination of IMC-A12 and CCI-779 (temsirolimus). (Phase II)

SECONDARY OBJECTIVES:

I. To determine the maximal percent decrease in PSA from baseline. II. To determine the change in PSA doubling time (PSADT). III. To determine the time to PSA progression and 6-month progression-free survival (PFS).

IV. To determine the rate of adverse events.

EXPLORATORY OBJECTIVES:

I. To evaluate changes in circulating tumor cell (CTC) numbers with time. II. To evaluate IGF1R and androgen receptor (AR) in CTCs and correlate with response.

III. To evaluate profiling CTCs at the molecular level by polymerase chain reaction (PCR) for prostate cancer-specific genes.

IV. To explore the association between clinical outcomes, administration of therapy, and serial fludeoxyglucose F 18 (FDG)-positron emission tomography (PET) imaging.

V. To correlate fluorine F 18 FMDHT (18-FDHT)-PET imaging findings with outcome measures of response.

VI. To perform tumor biopsies and evaluate biomarkers that may correlate with active feedback and tumor response to therapy, including anti-insulin receptor substrate 1 (IRS-1), anti-IRS-2, phosphorylated (p) protein kinase B (Akt)(S473), p-ribosomal protein S6 kinase (70/S6K), anti-phospho-AKT1 substrate 1 (proline-rich) (PRAS 40), and phosphatase and tensin homolog gene (PTEN) status.

OUTLINE: This is a multicenter study.

Patients receive cixutumumab intravenously (IV) over 60-70 minutes and temsirolimus IV over 30 minutes on days 1, 8, 15, and 22. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed adenocarcinoma of the prostate

  * Distant metastases evaluable by radionuclide bone scan, CT scan, or magnetic resonance imaging (MRI) within the past 28 days
* Evidence of progressive disease during androgen-deprivation therapy (including a trial of antiandrogen-withdrawal therapy), as defined by ≥ 1 of the following criteria:

  * Progressive measurable disease using conventional solid tumor criteria
  * Bone scan progression, defined as ≥ 2 new lesions on bone scan
  * Increasing PSA, defined as ≥ 2 consecutive rising PSA values over a reference value taken ≥ 1 week apart (the third PSA value must be greater than the second PSA value, if not, a fourth PSA value must be greater than the second PSA value)
* Castrate levels of serum testosterone (i.e., ≤ 50 ng/dL)
* No known brain metastases
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0-1 OR Karnofsky PS 70-100%
* Life expectancy > 6 months
* Leukocytes ≥ 3,000/μL
* Absolute neutrophil count (ANC) ≥ 1,500/μL
* Platelet count ≥ 100,000/μL
* Hemoglobin ≥ 9 g/dL
* Total bilirubin ≤ 2 times upper limit of normal (ULN)
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 2.5 times ULN
* Serum creatinine ≤ 1.5 times ULN
* Creatinine clearance ≥ 50 mL/min
* Able to adhere to the study visit schedule and other study requirements
* Fertile patients must use effective contraception before, during, and for 3 months after completion of study treatment
* Adequate lung function (pulmonary function test ≥ 70% for diffusion capacity of the lung for carbon monoxide [DLco])
* No poorly controlled diabetes mellitus

  * Patients with a history of diabetes are eligible provided their blood glucose is normal (i.e., fasting blood glucose < 120 mg/dL or < ULN) and they are on a stable dietary or therapeutic regimen
* No other malignancy within the past 3 years except for treated basal cell or squamous cell carcinoma of the skin or superficial transitional cell carcinoma of the bladder
* No uncontrolled major illness including, but not limited to, any of the following:

  * Active infection, including human immunodeficiency virus (HIV) infection or viral hepatitis
  * Symptomatic congestive heart failure (class III or IV)
  * Unstable angina pectoris
  * Myocardial infarction or acute coronary syndrome within the past year
  * Serious cardiac arrhythmia
  * Significant lung disease
  * Major psychiatric illness
* No other concurrent anticancer agents or treatments
* No prior chemotherapy, except for neoadjuvant chemotherapy
* No prior anti-insulin-like growth factor receptor (IGFR) agents or mammalian target of rapamycin (mTOR) inhibitors
* No prior strontium-89, rhenium-186, rhenium-188, or samarium-153 radionucleotide therapy
* Prior standard-dose radiotherapy to the pelvis for prostate cancer and/or additional external-beam radiotherapy to metastatic sites allowed
* More than 4 weeks since prior surgery, radiotherapy, combined androgen blockade (excluding single-agent gonadotropin releasing-hormone agonists/antagonists), or investigational therapies
* No concurrent second-line hormonal agents, including ketoconazole, diethylstilbestrol, other estrogen-like agents, or finasteride
* No concurrent corticosteroids unless patient is on a stable maintenance dose of hydrocortisone (≤ 30 mg/day) for ≥ 3 months

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2009-10; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dana Rathkopf, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (4):
- United States (4):
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - University of Wisconsin Hospital and Clinics, Madison, Wisconsin

RESULTS

PARTICIPANT FLOW:
Groups:
- IMC-A12: 6 mg/kg & Temsirolimus (CCI-779): 20 mg: Patients receive cixutumumab IV over 60-70 minutes and temsirolimus IV over 30 minutes on days 1, 8, 15, and 22. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Cixutumumab: Given IV
  Diagnostic Laboratory Biomarker Analysis: Correlative studies
  Temsirolimus: Given IV Arm -1 (Cycle=28 days, IMC-A12: 6 mg/kg IV over 60 min weekly, Temsirolimus (CCI-779): 20 mg IV over 30 min weekly)
- IMC-A12: 6 mg/kg & Temsirolimus (CCI-779): 25 mg: Patients receive cixutumumab IV over 60-70 minutes and temsirolimus IV over 30 minutes on days 1, 8, 15, and 22. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Cixutumumab: Given IV
  Diagnostic Laboratory Biomarker Analysis: Correlative studies
  Temsirolimus: Given IV Cycle=28 days, IMC-A12: 6 mg/kg IV over 60 min weekly, Temsirolimus (CCI-779): 25 mg IV over 30 min weekly
- IMC-A12: 20 mg/kg & Temsirolimus (CCI-779): 20 mg: Patients receive cixutumumab IV over 60-70 minutes and temsirolimus IV over 30 minutes on days 1, 8, 15, and 22. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Cixutumumab: Given IV
  Diagnostic Laboratory Biomarker Analysis: Correlative studies
  Temsirolimus: Given IV Cycle=21 days:IMC-A12: 20 mg/kg IV over 90 min on day 1 Temsirolimus (CCI-779): 20 mg IV over 30 min on day 1 Fluorine-18 2-Fluoro-2-deoxy-D-Glucose (18F-FDG): 10 mCi IVB at baseline, within 1 week of the 1st txt, 12 weeks, 24 weeks, and end of study
Period: Overall Study
Arm/Group | IMC-A12: 6 mg/kg & Temsirolimus (CCI-779): 20 mg | IMC-A12: 6 mg/kg & Temsirolimus (CCI-779): 25 mg | IMC-A12: 20 mg/kg & Temsirolimus (CCI-779): 20 mg
Started | 6 | 5 | 5
Completed | 6 | 5 | 5
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- IMC-A12: 6mg/kg Temsirolimus 20 mg: Patients receive cixutumumab IV over 60-70 minutes and temsirolimus IV over 30 minutes on days 1, 8, 15, and 22. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Cixutumumab: Given IV
  Diagnostic Laboratory Biomarker Analysis: Correlative studies
  Temsirolimus: Given IV Arm -1 (Cycle=28 days, IMC-A12: 6 mg/kg IV over 60 min weekly, Temsirolimus (CCI-779): 20 mg IV over 30 min weekly)
- IMC-A12: 6 mg/kg Temsirolimus 25 mg: Patients receive cixutumumab IV over 60-70 minutes and temsirolimus IV over 30 minutes on days 1, 8, 15, and 22. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Cixutumumab: Given IV
  Diagnostic Laboratory Biomarker Analysis: Correlative studies
  Temsirolimus: Given IV Cycle=28 days, IMC-A12: 6 mg/kg IV over 60 min weekly, Temsirolimus (CCI-779): 25 mg IV over 30 min weekly
- IMC-A12: 20 mg/kg Temsirolimus 20 mg: Patients receive cixutumumab IV over 60-70 minutes and temsirolimus IV over 30 minutes on days 1, 8, 15, and 22. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Cixutumumab: Given IV
  Diagnostic Laboratory Biomarker Analysis: Correlative studies
  Temsirolimus: Given IV Cycle=21 days:IMC-A12: 20 mg/kg IV over 90 min on day 1 Temsirolimus (CCI-779): 20 mg IV over 30 min on day 1 Fluorine-18 2-Fluoro-2-deoxy-D-Glucose (18F-FDG): 10 mCi IVB at baseline, within 1 week of the 1st txt, 12 weeks, 24 weeks, and end of study
- Total: Total of all reporting groups
Arm/Group | IMC-A12: 6mg/kg Temsirolimus 20 mg | IMC-A12: 6 mg/kg Temsirolimus 25 mg | IMC-A12: 20 mg/kg Temsirolimus 20 mg | Total
Number analyzed (Participants) | 6 | 5 | 5 | 16
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 0 | 2 | 2 | 4
  >=65 years | 6 | 3 | 3 | 12
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0
  Male | 6 | 5 | 5 | 16
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 1 | 0 | 1
  White | 6 | 4 | 5 | 15
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 6 | 5 | 5 | 16

OUTCOME MEASURES:

1. Primary Outcome: cTTP
Description: Defined as the time from the first day of treatment to the earliest one of the following: tumor progression by RECIST; unequivocal evidence of progression by bone scan (at least two new lesions with confirmation at subsequent imaging); new skeletal events; symptomatic progression; or other clinical events attributable to prostate cancer that necessitate major interventions.
  This Outcome Measure is related to the Phase II portion of the Trial, which did not occur.
  Therefore, there is no data to report.
Time Frame: Up to 4 weeks after completion of study treatment
Population: All patients had withdrawn from study prior to data analysis. This Outcome Measure is related to the Phase II portion of the Trial, which did not occur.
  Therefore, there is no data to report.
Groups:
- IMC-A12: 6 mg/kg Temsirolimus 20 mg: Patients receive cixutumumab IV over 60-70 minutes and temsirolimus IV over 30 minutes on days 1, 8, 15, and 22. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Cixutumumab: Given IV
  Diagnostic Laboratory Biomarker Analysis: Correlative studies
  Temsirolimus: Given IV Arm -1 (Cycle=28 days, IMC-A12: 6 mg/kg IV over 60 min weekly, Temsirolimus (CCI-779): 20 mg IV over 30 min weekly)
Arm/Group | IMC-A12: 6 mg/kg Temsirolimus 20 mg | IMC-A12: 6 mg/kg Temsirolimus 25 mg | IMC-A12: 20 mg/kg Temsirolimus 20 mg
Number analyzed (Participants) | 0 | 0 | 0

2. Primary Outcome: Tumor Response Rate
Description: Defined by modified Response Evaluation Criteria in Solid Tumors (RECIST) and/or the proportion of patients who achieve a greater than 50% reduction in serum PSA compared to baseline.
Time Frame: Up to 4 weeks after completion of study treatment
Measure: Count of Participants; unit: Participants
Arm/Group | IMC-A12: 6 mg/kg Temsirolimus 20 mg | IMC-A12: 6 mg/kg Temsirolimus 25 mg | IMC-A12: 20 mg/kg Temsirolimus 20 mg
Number analyzed (Participants) | 6 | 5 | 5
Participants
  Stable Disease | 2 | 4 | 1
  Progression of Disease | 4 | 1 | 4

3. Secondary Outcome: Change in PSA Doubling Time
Description: Compared using descriptive statistics. PSA doubling time is defined as the number of months it would take for PSA to increase two-fold. PSADT is inversely proportional to the slope of the regression line for the relation between log PSA and time. If this slope is negative, so the patient's PSA is going down over time, then the PSADT is negative.
Time Frame: Week 1, Week 5, Week 9, Week 13, Week 17, Week 21 and Week 25
Population: Outcome not calculated. PSA decline from baseline and imaging response (at twelve weeks) instead which are recognized PCWG3 endpoints for metastatic castration resistant disease was the outcome.
Arm/Group | IMC-A12: 6 mg/kg Temsirolimus 20 mg | IMC-A12: 6 mg/kg Temsirolimus 25 mg | IMC-A12: 20 mg/kg Temsirolimus 20 mg
Number analyzed (Participants) | 0 | 0 | 0

4. Secondary Outcome: Duration of Effect
Description: Summarized using descriptive statistics.
Time Frame: From the time of first dose until the time of progression, assessed up to 4 weeks after completion of study treatment
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | IMC-A12: 6 mg/kg Temsirolimus 20 mg | IMC-A12: 6 mg/kg Temsirolimus 25 mg | IMC-A12: 20 mg/kg Temsirolimus 20 mg
Number analyzed (Participants) | 6 | 5 | 5
weeks | 35 [10 to 60] | 17.5 [12 to 36] | 16 [4 to 22]

5. Secondary Outcome: Maximal Percentage Change in Serum PSA as Compared to Week 12 Versus Baseline
Description: Summarized using descriptive statistics (eg, mean, standard deviation, median, minimum, maximum).
  Maximum percent change in serum PSA (i.e., 100%*[(value at Week 12 minus value at baseline)/value at baseline])
Time Frame: From baseline to week 12
Measure: Median (95% Confidence Interval); unit: percentage change in Serum PSA
Arm/Group | IMC-A12: 6 mg/kg Temsirolimus 20 mg | IMC-A12: 6 mg/kg Temsirolimus 25 mg | IMC-A12: 20 mg/kg Temsirolimus 20 mg
Number analyzed (Participants) | 6 | 5 | 5
percentage change in Serum PSA | 8 [-47 to 63] | -1 [-29 to 26] | 203 [29 to 377]

6. Secondary Outcome: Progression-free Survival
Description: Summarized using descriptive statistics. Median PFS over time will be determined using Kaplan Meier method.
  This Outcome Measure was related to the Phase 2 portion of the study, which did not occur.
  Therefore, there is no data to report.
Time Frame: From the time of first dose until objective tumor progression or death, assessed up to 4 weeks after completion of study treatment
Population: All patients had withdrawn from study prior to data analysis.
Groups:
- Arm 1A: Patients receive cixutumumab IV over 60-70 minutes and temsirolimus IV over 30 minutes on days 1, 8, 15, and 22. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Cixutumumab: Given IV
  Diagnostic Laboratory Biomarker Analysis: Correlative studies
  Temsirolimus: Given IV Cycle=21 days:IMC-A12: 20 mg/kg IV over 90 min on day 1 Temsirolimus (CCI-779): 20 mg IV over 30 min on day 1 Fluorine-18 2-Fluoro-2-deoxy-D-Glucose (18F-FDG): 10 mCi IVB at baseline, within 1 week of the 1st txt, 12 weeks, 24 weeks, and end of study
Arm/Group | IMC-A12: 6 mg/kg Temsirolimus 20 mg | IMC-A12: 6 mg/kg Temsirolimus 25 mg | Arm 1A
Number analyzed (Participants) | 0 | 0 | 0

7. Secondary Outcome: Rate of Adverse Events According to NCI CTCAE Version 4.0
Description: Adverse event summaries will be organized by body system, frequency of occurrence, intensity (ie, severity grade), and causality or attribution.
  Please see Adverse Event/Serious Adverse Event Section.
Time Frame: Up to 4 weeks after completion of study treatment
Measure: Number; unit: percentage of participants affected
Arm/Group | IMC-A12: 6 mg/kg Temsirolimus 20 mg | IMC-A12: 6 mg/kg Temsirolimus 25 mg | IMC-A12: 20 mg/kg Temsirolimus 20 mg
Number analyzed (Participants) | 6 | 5 | 5
percentage of participants affected | 100 | 100 | 60

ADVERSE EVENTS:
Arm/Group | IMC-A12: 6mg/kg Temsirolimus 20 mg | IMC-A12: 6 mg/kg Temsirolimus 25 mg | IMC-A12: 20 mg/kg Temsirolimus 20 mg
Serious Adverse Events (participants affected / at risk) | 3/6 | 1/5 | 1/5
Other Adverse Events (participants affected / at risk) | 6/6 | 5/5 | 3/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IMC-A12: 6mg/kg Temsirolimus 20 mg (N=6) | IMC-A12: 6 mg/kg Temsirolimus 25 mg (N=5) | IMC-A12: 20 mg/kg Temsirolimus 20 mg (N=5)
Confusion (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Lipase increased (Investigations) | 2 (2) | 0 (0) | 0 (0)
Serum amylase increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Optic nerve disorder (Eye disorders) | 0 (0) | 0 (0) | 1 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IMC-A12: 6mg/kg Temsirolimus 20 mg (N=6) | IMC-A12: 6 mg/kg Temsirolimus 25 mg (N=5) | IMC-A12: 20 mg/kg Temsirolimus 20 mg (N=5)
Alkaline phosphatase increased (Investigations) | 1 (2) | 1 (6) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Cholesterol high (Investigations) | 0 (0) | 2 (2) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Fatigue (General disorders) | 2 (2) | 2 (3) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 1 (2) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 4 (36) | 3 (35) | 1 (3)
Hypertriglyceridemia (Metabolism and nutrition disorders) | 2 (6) | 2 (4) | 2 (2)
Hypophosphatemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Mucositis oral (Gastrointestinal disorders) | 1 (1) | 3 (5) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Neutrophil count decreased (Investigations) | 0 (0) | 1 (7) | 0 (0)
Peripheral motor neuropathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Platelet count decreased (Investigations) | 1 (3) | 0 (0) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Psychiatric disorders - Other, specify (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Rectal pain (Gastrointestinal disorders) | 0 (0) | 1 (2) | 0 (0)
Renal and urinary disorders - Other, specify (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Serum amylase increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Skin infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Thromboembolic event (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Tooth infection (Infections and infestations) | 1 (2) | 0 (0) | 0 (0)
Weight loss (Investigations) | 1 (1) | 1 (1) | 0 (0)
White blood cell decreased (Investigations) | 1 (1) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
cTTP This Outcome Measure is related to the Phase II portion of the Trial, which did not occur. All patients had withdrawn from study prior to data analysis. Therefore, there is no data to report for this measure.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less